CLINICAL TRIAL: NCT04295616
Title: The Additional Effect of Intrapulmonary Percussive Ventilation (IPV) on Respiration in People With Multiple Sclerosis (MS).
Brief Title: Additional Effect of Intrapulmonary Percussive Ventilation (IPV) on Respiration in People With Multiple Sclerosis (MS).
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 situation IPV is no longer allowed in the center
Sponsor: National Multiple Sclerosis Center (Other)
Collaborators: National MS Center Melsbroek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S 501553
Record Dates: First submitted 2020-02-11; First posted 2020-03-04 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPV & active breathing training (Experimental): Intrapulmonary Percussive Ventilation (IPV) and active breathing exercises, provided by trained speech and language therapists.
  This training will be performed in combination with a multidisciplinary rehabilitation programme.
  Interventions: Device: Intrapulmonary percussive ventilation (IPV); Behavioral: Active breathing training
- Active breathing training only (Active Comparator): Active breathing training provided by trained speech therapists. This training will be performed in combination with a multidisciplinary rehabilitation programme.
  Interventions: Behavioral: Active breathing training

INTERVENTIONS:
Device: Intrapulmonary percussive ventilation (IPV) — IPV is a well-tolerated method to pump air jets into the lungs via a mouth mask at frequencies of 100-400 pulses per minute.
  Each IPV session lasts 15 minutes, whereby the person with MS is firstly administered with a mask for 3 minutes at a high frequency (250 to 400 cycles per minute) and then 12 minutes with a low frequency (75 to 150 cycles per minute). The pressure (1.1 - 1.4 bar) is adjusted so that it is comfortable for every participant, yet there is the maximum possible expansion of the thorax. The sessions are given by speech therapists who are familiar with IPV. The IPV treatment will be provided 5 days a week, during 3 or 4 weeks.
  Arms: IPV & active breathing training
Behavioral: Active breathing training — The active breathing exercises are based on the flow-based incentive spirometer (Inspirix). The Inspirix is a device consisting of a tube with a ball. A plastic tube is connected to the device with a mouthpiece in which the person with MS will has to breathe in and out. The device is equipped with a control button to build up the resistance (number of cc / sec). The aim is to train the inspiratory and expiratory volume as well as the inspiratory and expiratory exhalation force. These exercises are offered 5 times a week in groups under the supervision of an experienced speech therapist, during 3 or 4 weeks.

SUMMARY:
This study aims to investigate whether intrapulmonary percussive ventilation (IPV) in combination with active breathing exercises using the flow-based incentive spirometer (Inspirix) has a positive effect on the respiratory values in people with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The primary research question includes "what is the additional effect of intensive IPV treatment in combination with active breathing exercises on respiratory power (Peak Expiratory Flow, PEF) in people with MS?".

In a single-center randomized clinical trial, 96 people with MS-related respiratory problems will be allocated to either the intervention group (IPV + active breathing training) or the control group (active breathing training only). Interventions will be provided by trained speech- and language therapists, in combination with a multidisciplinary rehabilitation programme of 3 weeks. Pre- en posttraining assessment includes measures of respiration, speech and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis MS
* inpatient in the National Multiple Sclerosis Center Melsbroek for at least 3 weeks in the period Jan-Dec 2020
* adequate lip closure
* adequate cognitive functioning (MMSE>26/30 & clinical observation)
* Peak Expiratory Flow (PEF) with a cut off score of 80% or lower

Exclusion Criteria:

* IPV or other breathing treatment of more than 1x/week within 3 months prior to study participation
* MS relapse within 3 months prior to study participation
* asthma or Chronic Obstructive Pulmonary Disease (COPD)
* infection of lower respiratory tract within 6 weeks prior to study participation
* infection of upper respiratory tract within 2 weeks prior to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Change in breathing force | pre- post (3 weeks) (some participants also at 4 weeks)
  Change in Peak Expiratory Flow (PEF)- Maximum flow achieved during a maximum forced exhalation.

SECONDARY OUTCOMES:
Change in Pulmonary Dysfunction Index (PDI) | pre- post (3 weeks) (some participants also at 4 weeks)
  To determine the PDI, the assessor judges the cough force and the ability of the person to count on 1 exhalation. PDI scores vary between 4 and 11 and a higher score indicates increasing respiratory difficulties.
Change in Maximum Phonation time (MFT) | pre- post (3 weeks) (some participants also at 4 weeks)
  The maximum phonation time (MFT) (in seconds) is measured at a comfortable pitch of the voice. The patient is instructed to breathe in as deeply as possible and to hold / a / as long as possible. MFT is measured three times and the longest value is retained.
Change in Voice Handicap Index (VHI-10) | pre- post (3 weeks) (some participants also at 4 weeks)
  The Voice Handicap Index (VHI-10) 10-item questionnaire assesses the psychosocial impact on the voice as perceived by the individual. The VHI-10 scores range from 0 to 40, with increasing scores indicating increased psychosocial impact. A score of 11 or higher implies a voice handicap.
Change in Vital Capacity (VC) | pre- post (3 weeks) (some participants also at 4 weeks)
  Maximum amount of air that is exhaled after a deep inhalation. The person is asked to breathe out as deeply as possible in the mouthpiece after a deep inhalation.
Change in Maximum Inspiratory Pressure (MIP) | pre- post (3 weeks) (some participants also at 4 weeks)
  Maximum inspiratory pressure at which the person inhales against a resistance.
Change in Maximum Expiratory Pressure (MEP) | pre- post (3 weeks) (some participants also at 4 weeks)
  MEP is the highest pressure that arises during a powerful exhalation against a resistance.
Change in Visual Analogue Scale (VAS) for fatigue | pre- post (3 weeks) (some participants also at 4 weeks)
  This is an assessment instrument consisting of a straight line of 10 cm with two opposite statements at both ends. On the left is the statement "not at all tired" and on the right "extremely tired".

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Noë, Msc, Principal Investigator — National MS Center Melsbroek - Speech and Language Therapy
Locations (1):
- National MS Center, Melsbroek, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National MS Center Melsbroek — https://mscenter.be/en